CLINICAL TRIAL: NCT06255678
Title: Angio-based Final Functional Effect of PCI (AFFE PCI): a Prospective Multi-center Study of Post-PCI vFFR Impact on Clinical Outcomes and Residual Angina
Brief Title: Angio-based Final Functional Effect of PCI
Acronym: AFFE-PCI
Status: Recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Mariusz Tomaniak, Tomaniak Mariusz MD PhD Assoc. Prof., Medical University of Warsaw
Other Study IDs: AFFE-PCI
Record Dates: First submitted 2024-01-16; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Acute Coronary Syndrome; Non ST Segment Elevation Acute Coronary Syndrome; Chronic Coronary Syndrome
Keywords: vFFR; ACS; NST-ACS; Angiography-based FFR; Quality of life; Residual angina
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing PCI: Assessment of ΔvFFR and vFFR after PCI and adverse clinical outcomes, residual angina and quality of life using the validated Seattle Angina Questionnaire (SAQ) and EuroQol 5-level 5-dimensional questionnaire (EQ-5D-5L) in patients with CCS or ACS.
  Interventions: Diagnostic Test: Angiography-based vessel fractional flow reserve (vFFR) calculation

INTERVENTIONS:
Diagnostic Test: Angiography-based vessel fractional flow reserve (vFFR) calculation — vFFR is calculated from routinely taken angiography images during PCI using a CAAS workstation (Pie Medical Imaging, Maastricht, the Netherlands)

SUMMARY:
Fractional flow reserve (FFR) has revolutionized the diagnosis and treatment of coronary artery disease (CAD), and more recently, post percutaneous coronary intervention (post-PCI) FFR has emerged as an independent predictor of cardiovascular events, enabling the identification of cases requiring additional optimization of the implanted stent. Modern technologies allow less invasive alternatives to traditional FFR measurement - angiography-based vessel fractional flow reserve (vFFR) and derivative ΔvFFR, which is calculated by a difference between the post-PCI vFFR and pre-PCI vFFR. In large clinical studies, the good accuracy between vFFR and FFR - measured before and after PCI - has been confirmed. However, insufficient data is available about the value of post-vFFR and ΔvFFR as prognostic values and indicators of patient health.

This is a prospective multicenter register study analyzing the association between the value of ΔvFFR, vFFR after PCI and adverse clinical outcomes, residual angina and quality of life using the validated Seattle Angina Questionnaire (SAQ) and EuroQol 5-level 5-dimensional questionnaire (EQ-5D-5L). Patients undergoing PCI for chronic coronary syndromes (CCS), non-ST-segment elevation acute coronary syndromes (NST-ACS) or ST-Segment Elevation Myocardial Infarction (STEMI) will be enrolled in this study.

DETAILED DESCRIPTION:
The primary goal of this prospective multicenter register study is to evaluate the association between the value of vFFR after PCI and adverse clinical outcomes, residual angina and quality of life using the validated Seattle Angina Questionnaire (SAQ) and EuroQol 5-level 5-dimensional questionnaire (EQ-5D-5L) at 6 and 24 months following PCI. The primary composite endpoint is defined as a major adverse cardiovascular event (MACE) including all-cause death, target-vessel myocardial infarction (TVMI), and target vessel revascularization (TVR)] at 6, 12 and 24-month follow-ups. Patients undergoing PCI for chronic coronary syndromes (CCS), non-ST-segment elevation acute coronary syndromes (NST-ACS) or or ST-Segment Elevation Myocardial Infarction (STEMI) will be enrolled in this study. The analyses of the primary endpoint will be stratified according to the following subgroups:

* Diabetes/non-diabetes
* Glomerular filtration rate (GFR)≥60/GFR<60 [ml/min./1,73m2]
* Focal/diffuse atherosclerosis
* Multivessel/single-vessel disease
* CCS/NST-ACS/STEMI
* CCS/ACS

The patients' coronary angiograms will be analyzed using a CAAS workstation (Pie Medical Imaging, Maastricht, the Netherlands) enrolled at the Invasive Cardiology Unit of the 1st Department of Cardiology, Medical University of Warsaw (Poland) and other centers in Poland.

ELIGIBILITY:
Inclusion Criteria:

* Percutaneous coronary intervention (PCI) for chronic coronary syndromes (CCS) or acute coronary syndromes (ACS)
* Adequate quality of angiogram enabling vFFR analysis (available two angiographic views with ≥30° differences in rotation/angulation, the possibility of vessel contour selection, proper quality of the images, vessels without severe overlapping, tortuosity, foreshortening and poor vessel opacification)
* Age >18 years
* The patient's written informed consent has been obtained before the procedure

Exclusion Criteria:

* Cardiogenic shock, pulmonary oedema
* Severe hemodynamical instability
* Prior coronary artery bypass grafting (CABG)
* Active bleeding
* Acute and chronic inflammatory conditions
* Acute mechanical complications of myocardial infarction
* Congenital heart disease
* Heart transplantation
* Non-cardiac comorbidities with a life expectancy of less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with percutaneous coronary intervention (PCI) for chronic coronary syndromes (CCS) or acute coronary syndromes (ACS)
Sampling Method: Non-Probability Sample
Enrollment: 2005 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of MACE defined as all-cause death, target-vessel myocardial infarction (TVMI) and target vessel revascularization (TVR). | 24 months

SECONDARY OUTCOMES:
Rate of MACE defined as all-cause death, target-vessel myocardial infarction (TVMI) and target vessel revascularization (TVR). | 6 months, 12 months
Rate of all-cause death | 6 months, 12 months, 24 months
Rate of target-vessel myocardial infarction (TVMI) | 6 months, 12 months, 24 months
Rate of target-vessel target vessel revascularization (TVR) | 6 months, 12 months, 24 months
Symptoms of angina and quality of life assessed by the score of EuroQol 5-level 5-dimensional questionnaire (EQ-5D-5L) | 6 months, 12 months, 24 months
  The EQ-5D-5L scale asses the patient's self-rated health in five categories (each category 1-5) - higher values indicate worse performance. Additionally, the patient fulfill vertical visual analog scale from 0 to 100, where higher scores indicate better function.
Symptoms of angina and quality of life assessed by score of the Seattle Angina Questionnaire (SAQ) | 6 months, 12 months, 24 months
  The SAQ provides results for 6 categories. The patient can receive between 0 and 100 points in each category, where 100 represents the best score.
Correlation of post-percutaneous coronary intervention (PCI) vessel fractional flow reserve (vFFR) with score of Seattle Angina Questionnaire (SAQ). | 6 months, 12 months, 24 months
  The SAQ provides results for 6 categories. The patient can receive between 0 and 100 points in each category, where 100 represents the best score. vFFR values are within the range 0-1, where higher values indicate better function.
Correlation of ΔvFFR with score of Seattle Angina Questionnaire (SAQ). | 6 months, 12 months, 24 months
  The SAQ provides results for 6 categories. The patient can receive between 0 and 100 points in each category, where 100 represents the best score.
Correlation of post-percutaneous coronary intervention (PCI) vessel fractional flow reserve (vFFR) with score of EuroQol 5-level 5-dimensional questionnaire (EQ-5D-5L). | 6 months, 12 months, 24 months
  The EQ-5D-5L scale asses the patient's self-rated health in five categories (each category 1-5) - higher values indicate worse performance. Additionally, the patient fulfill vertical visual analog scale from 0 to 100, where higher scores indicate better function. vFFR values are within the range 0-1, where higher values indicate better function.
Correlation of ΔvFFR with score of EuroQol 5-level 5-dimensional questionnaire (EQ-5D-5L). | 6 months, 12 months, 24 months
  The EQ-5D-5L scale asses the patient's self-rated health in five categories (each category 1-5) - higher values indicate worse performance. Additionally, the patient fulfill vertical visual analog scale from 0 to 100, where higher scores indicate better function.
AUC for the optimal cutoff point for post-percutaneous coronary intervention (PCI) vessel fractional flow reserve (vFFR) for significant prediction of MACE | 6 months, 12 months, 24 months
  MACE defined as all-cause death, target-vessel myocardial infarction (TVMI) and target vessel revascularization (TVR).
AUC for the optimal cutoff point for ΔvFFR useful for prediction of MACE | 6 months, 12 months, 24 months
  MACE defined as all-cause death, target-vessel myocardial infarction (TVMI) and target vessel revascularization (TVR).
AUC for the optimal cutoff point for post-percutaneous coronary intervention (PCI) vessel fractional flow reserve (vFFR) useful for prediction of higher than median SAQ score. | 6 months, 12 months, 24 months
  The SAQ provides results for 6 categories. The patient can receive between 0 and 100 points in each category, where 100 represents the best score. vFFR values are within the range 0-1, where higher values indicate better function.
AUC for the optimal cutoff point for post-percutaneous coronary intervention (PCI) vessel fractional flow reserve (vFFR) useful for prediction of higher than median EQ-5D-5L score. | 6 months, 12 months, 24 months
  The scale asses the patient's self-rated health in five categories (each category 1-5) - higher values indicate worse performance. Additionally, the patient fulfill vertical visual analog scale from 0 to 100, where higher scores indicate better function. vFFR values are within the range 0-1, where higher values indicate better function.
AUC for the optimal cutoff point for ΔvFFR useful for prediction of higher than median SAQ score. | 6 months, 12 months, 24 months
  The SAQ provides results for 6 categories. The patient can receive between 0 and 100 points in each category, where 100 represents the best score.
AUC for the optimal cutoff point for ΔvFFR useful for prediction of higher than median EQ-5D-5L score. | 6 months, 12 months, 24 months
  The scale asses the patient's self-rated health in five categories (each category 1-5) - higher values indicate worse performance. Additionally, the patient fulfill vertical visual analog scale from 0 to 100, where higher scores indicate better function.
Rate of revascularization of any vessel due to exacerbation of angina symptoms. | 6 months, 12 months, 24 months
  Decisions on the performance of revascularization will be made by the attending physician according to the clinical features and available methods.
Rate of definite and probable stent thrombosis. | 6 months, 12 months, 24 months
Rate of clinically driven invasive coronary angiography due to exacerbation of angina symptoms. | 6 months, 12 months, 24 months
  Decisions on the performance of invasive coronary angiography will be made by the attending physician according to the clinical features.
AUC for the value of in-stent vFFR gradient in predicting the rate of MACE | 6 months, 12 months, 24 months
  vFFR values are within the range 0-1, where higher values indicate better function.
AUC for the value of 3-vessel post-PCI vFFR burden (sum of the vFFR estimated in the three main epicardial arteries) in predicting the rate of MACE | 6 months, 12 months, 24 months
  3-vessel post-PCI vFFR will be defined as the sum of the post-PCI vFFR values derived for each vessel (left anterior descending, circumflex, right coronary artery).

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided